CLINICAL TRIAL: NCT04967794
Title: Effectiveness of Teleorientation in Oral Hygiene During the COVID-19 Pandemic, a Randomized Clinical Trial
Brief Title: Effectiveness of Teleorientation in Oral Hygiene During the COVID-19 Pandemic
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Marília Goulardins, Master's student in Pediatric Dentistry, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CAAE 39685920.7.0000.5419
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Dental Caries in Children
Keywords: eHealth, mobile health

STUDY DESIGN:
Intervention Model Description: The study population will be divided into three groups that will receive the intervention by communication platform, teleconsultation platform in health and in person.all individuals participating in the group will receive toothbrushing guidelines as a preventive measure for the development of dental caries
Who Masked: Participant
Masking Description: The clinical trial is a simple blind study in which the sample will be randomized into three groups, whose participants will be "blinded" to the types of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Whatsapp (Active Comparator): Will receive standardized brushing Teleorientation consultation through the Whatsapp communication platform
  Interventions: Other: Teleorientation and Tooth Brushing Orientation
- Group Vídeo for Health (Active Comparator): You will receive a standardized brushing Teleorientation consultation through the V4H Platform, created specifically for Teleconsultations
  Interventions: Other: Teleorientation and Tooth Brushing Orientation
- Group de Orientação presencial (Active Comparator): You will receive a standardized face-to-face brushing orientation consultation.
  Interventions: Other: Teleorientation and Tooth Brushing Orientation

INTERVENTIONS:
Other: Teleorientation and Tooth Brushing Orientation — Guide children in toothbrushing with a preventive purpose during the COVID-19 pandemic

SUMMARY:
The present study aims to evaluate the effectiveness of Teleorientation in oral hygiene during Pandemic by COVID-19 in children aged 6 to 10 years, attended at the Pediatric Clinic of Forp. For this, a randomized clinical study will be carried out with the factor to be analyzed the comparison between synchronous and asynchronous teleorientation, the effectiveness of the transfer of knowledge in oral hygiene through video modeling and remote guidance. The response variables will be the assimilation of oral hygiene guidance through video modeling and synchronous guidance, the hypothesis is that educational content will have beneficial effects on children's oral health.

DETAILED DESCRIPTION:
This is a randomized clinical trial, whose sample is composed of thirty children aged 6 to 10 years, attended between the year 2019 and the beginning of 2020. The sample will be randomly randomized into 3 groups who received guidance on toothbrushing. group 1 will be done Teleorientation of tooth brushing through video call by the Whatsapp application, in group 2 will be done Teleorientation of toothbrushing through a platform designed exclusively for teleconsultations and group 3 will receive the same in-person brushing orientation.

The main purpose of the clinical trial is to develop and analyze a program of Teleorientation of Toothbrushing in children of the Pediatric Dentistry clinic of FORP.

The Specific Objectives are assess whether oral hygiene is taking place properly during the COVID-19 Pandemic, assess, through a questionnaire, the level of understanding of parents and caregivers regarding the information received. This project will be designed as a randomized study with a two-month follow-up. The study factor will be to compare synchronous with asynchronous teleorientation, the effectiveness of knowledge transfer in oral hygiene through video modeling and remote orientation. The response variables will be the assimilation of guidance in oral hygiene by video modeling and by synchronous guidance, the hypothesis is that educational content will have beneficial effects on the oral health of children. The procedures will be performed at the Pediatric Dentistry Clinic of the Faculty of Dentistry of Ribeirão Preto - University of São Paulo - FORP/USP. The CONSORT guide (Schulz et al., 2010) for randomized controlled trials will be followed for the design of the present study.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6 to 8 years old,
* attended at Forp's Pediatric Dentistry Clinic,
* with complete record in the medical record,
* parents or caregivers who have Smartphone and Internet access
* and who are willing to download the V4H and
* WhatsApp application and
* accept to participate in all stages of the research upon acceptance of the consent form.

Exclusion Criteria

* :Children who present pain and/or spontaneous sensitivity,
* motor difficulties and
* health disorders .

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Estimated)

PRIMARY OUTCOMES:
Individual assessment of groups | 1 month
  Assess the children's visible plaque index individually by photo

CONTACTS AND LOCATIONS:
Locations (1):
- Marilia G Gomes, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Make the study visible to other researchers through the sharing link

REFERENCES:
- [Background] Lotto M, Strieder AP, Ayala Aguirre PE, Oliveira TM, Andrade Moreira Machado MA, Rios D, Cruvinel T. Parental-oriented educational mobile messages to aid in the control of early childhood caries in low socioeconomic children: A randomized controlled trial. J Dent. 2020 Oct;101:103456. doi: 10.1016/j.jdent.2020.103456. Epub 2020 Aug 20. PMID 32827598
- Available data/document: Informed Consent Form: CAAE 39685920.7.0000.5419 — https://plataformabrasil.saude.gov.br/ — Through this address it is possible to identify the information about acceptance by the ethics committee of Univerdade São Paulo and also the consent form